CLINICAL TRIAL: NCT03938857
Title: DEXMEDETOMIDINE OPIOID SPARING EFFECT IN MECHANICALLY VENTILATED CHILDREN: Phase 1b, Multicenter, Double Blind Randomized Controlled Dose Escalating Trial of Fentanyl vs. Fentanyl + Dexmedetomidine as the Initial Regimen for Maintenance of Sedation in Mechanically-ventilated, Critically Ill Children
Brief Title: DOSE Trial of Opioid Sparing Effect
Acronym: DOSE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment challenging during the pandemic COVID 19
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Johns Hopkins University (Other); Intermountain Health Care, Inc. (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00102267; 5U24TR001608 (NIH)
Record Dates: First submitted 2019-04-25; First posted 2019-05-06 (Actual); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Dexmedetomidine; Mechanical Ventilation Complication; Critically Ill
MeSH Terms: conditions — Critical Illness | interventions — Fentanyl; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Phase 1b randomized, double-blind, placebo-controlled dose escalation trial. The study will randomize participants to receive placebo (fentanyl standard of care) titrated to sedation+saline placebo (bolus+infusion) or one of the following 3 Dexmedetomidine treatment arms in a sequential cohort fashion: Cohort 1: Fentanyl SOC titrated to sedation + Dexmedetomidine (0.5mcg/kg bolus load + 0.2 mcg/kg/hr infusion); Cohort 2: Fentanyl SOC titrated to sedation + Dexmedetomidine (0.5mcg/kg bolus load + 0.5mcg/kg/hr infusion); Cohort 3: Fentanyl SOC titrated to sedation + Dexmedetomidine (0.5mcg/kg bolus load + 0.7mcg/kg/hr infusion).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Fen. SOC+saline placebo (bolus+infusion) (Placebo Comparator): Fentanyl standard of care (SOC) titrated to sedation + saline placebo (bolus + infusion)
  Interventions: Drug: Fentanyl
- Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) (Active Comparator): Fentanyl SOC titrated to sedation + Dexmedetomidine (0.5mcg/kg bolus load + 0.2mcg/kg/hr infusion)
  Interventions: Drug: Fentanyl; Drug: Dexmedetomidine
- Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) (Active Comparator): Fentanyl SOC titrated to sedation + Dexmedetomidine (0.5mcg/kg bolus load + 0.5mcg/kg/hr infusion)
  Interventions: Drug: Fentanyl; Drug: Dexmedetomidine
- Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr) (Active Comparator): Fentanyl SOC titrated to sedation + Dexmedetomidine (0.5mcg/kg bolus load + 0.7mcg/kg/hr infusion)
  Interventions: Drug: Fentanyl; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Fentanyl — Fentanyl standard of care
Drug: Dexmedetomidine — Dexmedetomidine (0.5 mcg/kg + 0.2 mcg/kg/hr)
  Arms: Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr)
Drug: Dexmedetomidine — Dexmedetomidine (0.5 mcg/kg + 0.5 mcg/kg/hr)
  Arms: Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr)
Drug: Dexmedetomidine — Dexmedetomidine (0.5 mcg/kg + 0.7 mcg/kg/hr)
  Arms: Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)

SUMMARY:
Multicenter, double blind randomized controlled trial of fentanyl vs. fentanyl + dexmedetomidine as the initial regimen for maintenance of sedation in mechanically-ventilated, critically ill children.

This trial will evaluate the opioid-sparing effect of dexmedetomidine when administered with fentanyl to mechanically ventilated, critically ill children. Study drug or placebo will be administered with fentanyl, which will be titrated to achieve sedation scores consistent with response to light touch. Plasma samples and bedside assessments for pain, sedation, and delirium will be collected.

DETAILED DESCRIPTION:
Phase 1b randomized, double-blind, placebo-controlled dose escalation trial of sedation regimens in critically ill children. Testing the hypothesis of mean daily fentanyl dose through day 7 of mechanical ventilation will be reduced by ≥25% by the addition of dexmedetomidine to fentanyl therapy. This trial will involve multiple clinical sites. Randomization will occur by individual and investigators will be blinded to study/treatment arm. The statistical analysis will account for center effects, participant characteristics (including post-surgical state), and changes over time to minimize bias. In addition, PIs and study coordinators will undergo training to standardize assessment procedures. The study will randomize participants to receive placebo (fentanyl standard of care) titrated to sedation+saline placebo (bolus+infusion) or one of the following 3 Dexmedetomidine treatment arms in a sequential cohort fashion: Cohort 1: Fentanyl SOC titrated to sedation + Dexmedetomidine (0.5mcg/kg bolus load + 0.2 mcg/kg/hr infusion); Cohort 2: Fentanyl SOC titrated to sedation + Dexmedetomidine (0.5mcg/kg bolus load + 0.5mcg/kg/hr infusion); and, Cohort 3: Fentanyl SOC titrated to sedation + Dexmedetomidine (0.5mcg/kg bolus load + 0.7mcg/kg/hr infusion).

An interim analysis is planned for this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 0 to <18 years at the time of enrollment.
2. If < 6 months postnatal age, gestational age ≥ 35 weeks.
3. Admitted to an intensive care unit.
4. Planned or anticipated mechanically ventilation for ≥2 days.
5. Require sedation to maintain mechanical ventilation per clinical judgment.
6. No contraindication to receipt of fentanyl or dexmedetomidine per clinician judgment.
7. Availability and willingness of the parent/legal guardian to provide written informed consent.

Exclusion Criteria:

1. Previous participation in this study.
2. Severe traumatic brain injury as the underlying etiology for critical illness requiring mechanical ventilation or baseline pediatric cerebral performance category (PCPC) >3.
3. Planned receipt of sedatives other than fentanyl or dexmedetomidine.
4. Anticipated receipt of neuromuscular blockade for >48 consecutive hours during the study period.
5. Receipt of fentanyl or dexmedetomidine via continuous infusion for >12 hours in the 24 hours prior to enrollment.
6. Extracorporeal life support (including renal replacement therapy, extracorporeal membrane oxygenation, ventricular assist device, etc.) at the time of enrollment.
7. Chronic use of or recent overdose of serotonergic agents (selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), monoamine oxidase (MAO) inhibitors, cyclic antidepressants)
8. Known pregnancy
9. Known liver dysfunction, defined as: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2x the upper limit of normal for age
10. Known or impending renal failure defined as: anuria > or equal to 12 hours prior to enrollment or requiring renal replacement therapy
11. High risk children, define as: a. known heart block b. known bradyarrythmia including clinically significant bradycardia (defined as requiring chronotropic agents or cardiac pacing to treat)
12. Receipt of mechanical ventilation during an admission for cardiac surgery

Note: receipt of drugs other than fentanyl or dexmedetomidine for intubation, and receipt of neuromuscular blockage for intubation, will not be considered exclusionary criteria.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Benjamin, MD, Principal Investigator — Duke Clinical Research Institute
Locations (19):
- United States (19):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Florida, Shands Children's Hospital, Gainesville, Florida
  - Indiana University Health, Riley Hospital for Children, Indianapolis, Indiana
  - Our Lady of the Lake Children's Hospital, Baton Rouge, Louisiana
  - UMass Memorial Medical Center, Children's Center, Worcester, Massachusetts
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Saint Louis University, Cardinal Glennon Children's Hospital, St Louis, Missouri
  - University of New Mexico Children's Hospital, Albuquerque, New Mexico
  - University of Buffalo, Oishei Children's Hospital, Buffalo, New York
  - University of Rochester Medical Center, Golisano Children's Hospital, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Rainbow Babies and Children's Hospital, University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - MetroHealth System, Case CTSA, Cleveland, Ohio
  - Oregon Health and Science University, Doernbecher Children's Hospital, Portland, Oregon
  - Drexel University, St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Medical University of South Carolina Children's Hospital, Charleston, South Carolina
  - University of Texas - Health Science Center San Antonio, San Antonio, Texas
  - Primary Children's Medical Center- University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boutzoukas AE, Olson R, Sellers MA, Fischer G, Hornik CD, Alibrahim O, Iheagwara K, Abulebda K, Bass AL, Irby K, Subbaswamy A, Zivick EE, Sweney J, Stormorken AG, Barker EE, Lutfi R, McCrory MC, Costello JM, Ackerman KG, Munoz Pareja JC, Dean JM, Abdelsamad N, Hanley DF Jr, Mould WA, Lane K, Stroud M, Feger BJ, Greenberg RG, Smith PB, Benjamin DK Jr, Hornik CP, Zimmerman KO, Becker ML. Mechanisms to expedite pediatric clinical trial site activation: The DOSE trial experience. Contemp Clin Trials. 2023 Feb;125:107067. doi: 10.1016/j.cct.2022.107067. Epub 2022 Dec 25. PMID 36577492

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled were in a pediatric intensive care setting, critically ill and requiring ventilatory support and pain management associated with such.
Period: Overall Study
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Started | 6 | 12 | 12 | 0
Completed | 5 | 12 | 12 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was prematurely terminated and no participants were enrolled in the Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr) group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr) | Total
Number analyzed (Participants) | 6 | 12 | 12 | 0 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.8 (6.8) | 2.5 (2.8) | 2.6 (3.7) |  | 2.8 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 4 |  | 12
  Male | 3 | 7 | 8 |  | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 |  | 2
  Not Hispanic or Latino | 5 | 11 | 10 |  | 26
  Unknown or Not Reported | 1 | 0 | 1 |  | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  | 0
  Asian | 0 | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0
  Black or African American | 3 | 3 | 1 |  | 7
  White | 3 | 8 | 8 |  | 19
  More than one race | 0 | 0 | 1 |  | 1
  Unknown or Not Reported | 0 | 1 | 2 |  | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 12 | 12 |  | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Daily Dose of Fentanyl in mcg/kg/hr (Micrograms Per Kilogram Per Hour)
Description: Characterize the opioid-sparing effect of dexmedetomidine when co-administered with fentanyl in children receiving mechanical ventilation. Characterization of differences between dosing exposures for the four groups will allow estimation of the opioid-sparing effect of dexmedetomidine.
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Population: Patients who did not have fentanyl reported were excluded. No participants were enrolled in the Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr) group.
Measure: Mean (Standard Deviation); unit: mcg/kg/hr
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 6 | 12 | 12 | 0
mcg/kg/hr | 2.25 (2.15) | 2.68 (1.53) | 3.23 (3.30) |
Statistical Analysis 1: Comparison: Fen. SOC+Saline Placebo (Bolus+Infusion) vs Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) vs Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr); Placebo group compared to combined Dexmedetomidine groups; Test type: Other; p = 0.814, Mixed Models Analysis; Slope = -0.1088295, 95% CI 2-sided [-1.035508 to 0.8178494], Standard Error of Mean 0.4728041 — Estimated value represents interaction between treatment and days

2. Secondary Outcome: Sedation Based on the State Behavior Scale (SBS) Relative to Fentanyl Plasma Concentrations (Cmax)
Description: Characterize the exposure response relationships of fentanyl and dexmedetomidine when administered alone or in combination in children receiving mechanical ventilation. PK is known to be altered in children compared to adults, and in those with critical illness. Characterization of pharmacokinetic-pharmacodynamic relationships can improve dose optimization when dose may not be equivalent to plasma exposure and related effect. The SBS is a 6-point scale that ranges from +2 to -3 with -3. Scores that are more negative reflect a more sedated state (-3). Scores that are more positive reflect a more agitated state (+2). Zero is awake and easily calmed.
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Population: Data not collected. The study was terminated early due to enrollment challenges.
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Sedation Based on SBS Scale Relative to Fentanyl Plasma Concentrations (Cmin)
Description: as for outcome 2
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Population: Data not collected. The study was terminated early due to enrollment challenges.
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Sedation Based on SBS Scale Relative to Fentanyl Plasma Concentrations (Css)
Description: as for outcome 2
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Population: Data not collected. The study was terminated early due to enrollment challenges.
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Sedation Based on SBS Scale Relative to Fentanyl Plasma Concentrations (AUC)
Description: as for outcome 2
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Population: Data not collected. The study was terminated early due to enrollment challenges.
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Sedation Based on SBS Scale Relative to Dexmedetomidine Plasma Concentrations (Cmax)
Description: as for outcome 2
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Population: Data not collected. The study was terminated early due to enrollment challenges.
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Sedation Based on SBS Scale Relative to Dexmedetomidine Plasma Concentrations (Cmin)
Description: as for outcome 2
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Population: Data not collected. The study was terminated early due to enrollment challenges.
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Sedation Based on SBS Scale Relative to Dexmedetomidine Plasma Concentrations (Css)
Description: as for outcome 2
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Population: Data not collected. The study was terminated early due to enrollment challenges.
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Sedation Based on SBS Scale Relative to Dexmedetomidine Plasma Concentrations (AUC)
Description: as for outcome 2
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Population: Data not collected. The study was terminated early due to enrollment challenges.
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Sedation Based on Richmond Agitation and Sedation Scale (RASS) Scale Relative to Fentanyl Plasma Concentrations (Cmax)
Description: Characterize the exposure response relationships of fentanyl and dexmedetomidine when administered alone or in combination in children receiving mechanical ventilation. PK is known to be altered in children compared to adults, and in those with critical illness. Characterization of pharmacokinetic-pharmacodynamic relationships can improve dose optimization when dose may not be equivalent to plasma exposure and related effect. The RASS is a 10-point scale that ranges from -5 to +4 with -5=unarousable and +4=combative. Zero means the patient is alert and calm.
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Population: Data not collected. The study was terminated early due to enrollment challenges.
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Sedation Based on RASS Scale Relative to Fentanyl Plasma Concentrations (Cmin)
Description: Characterize the exposure response relationships of fentanyl and dexmedetomidine when administered alone or in combination in children receiving mechanical ventilation. PK is known to be altered in children compared to adults, and in those with critical illness. Characterization of pharmacokinetic-pharmacodynamic relationships can improve dose optimization when dose may not be equivalent to plasma exposure and related effect. The RASS scale is a 10-pint scale that ranges from -5 to +4 with -5=unarousable and +4=combative. Zero means the patient is alert and calm.
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Population: Data not collected. The study was terminated early due to enrollment challenges.
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Sedation Based on RASS Scale Relative to Fentanyl Plasma Concentrations (Css)
Description: Characterize the exposure response relationships of fentanyl and dexmedetomidine when administered alone or in combination in children receiving mechanical ventilation. PK is known to be altered in children compared to adults, and in those with critical illness. Characterization of pharmacokinetic-pharmacodynamic relationships can improve dose optimization when dose may not be equivalent to plasma exposure and related effect. The RASS scale is a 10-point scale that ranges from -5 to +4 with -5=unarousable and +4=combative. Zero means the patient is alert and calm.
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Population: Data not collected. The study was terminated early due to enrollment challenges.
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Sedation Based on RASS Scale Relative to Fentanyl Plasma Concentrations (AUC)
Description: as for outcome 12
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Population: Data not collected. The study was terminated early due to enrollment challenges.
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Sedation Based on RASS Scale Relative to Dexmedetomidine Plasma Concentrations (Cmax)
Description: as for outcome 12
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Population: Data not collected. The study was terminated early due to enrollment challenges.
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Sedation Based on RASS Scale Relative to Dexmedetomidine Plasma Concentrations (Cmin)
Description: as for outcome 12
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Population: Data not collected. The study was terminated early due to enrollment challenges.
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Sedation Based on RASS Scale Relative to Dexmedetomidine Plasma Concentrations (Css)
Description: as for outcome 12
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Population: Data not collected. The study was terminated early due to enrollment challenges.
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Sedation Based on RASS Scale Relative to Dexmedetomidine Plasma Concentrations (AUC)
Description: as for outcome 12
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Population: Data not collected. The study was terminated early due to enrollment challenges.
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants Experiencing a Clinically Significant Episode of Hypotension
Description: Characterize the safety profile of fentanyl and dexmedetomidine when administered alone or in combination to children receiving mechanical ventilation.
Time Frame: up to 28 days or until discharge from the ICU (whichever is first)
Population: Participants with data collected. No participants were enrolled in the Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr) group.
Measure: Count of Participants; unit: Participants
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 5 | 12 | 12 | 0
Participants | 2 | 5 | 3 |

19. Secondary Outcome: Number of Participants Experiencing SAEs (Serious Adverse Events)
Time Frame: up to 28 days or until discharge from the ICU (whichever is first)
Population: No participants were enrolled in the Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr) group.
Measure: Count of Participants; unit: Participants
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 6 | 12 | 12 | 0
Participants | 0 | 2 | 1 |

20. Secondary Outcome: Mean Number of SAEs (Serious Adverse Events) Experienced by Participants
Time Frame: up to 28 days or until discharge from the ICU (whichever is first)
Population: Participants who experienced at least one SAE. No participants were enrolled in the Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr) group.
Measure: Mean (Standard Deviation); unit: serious adverse events
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 0 | 2 | 1 | 0
serious adverse events |  | 1 (0) | 1 (NA) — Only one participant experienced an SAE. |

21. Secondary Outcome: Number of Participants Experiencing a Clinically Significant Episode of Bradycardia
Description: as for outcome 18
Time Frame: up to 28 days or until discharge from the ICU (whichever is first)
Population: Participants with data collected. No participants were enrolled in the Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr) group.
Measure: Count of Participants; unit: Participants
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 5 | 12 | 12 | 0
Participants | 2 | 3 | 1 |

22. Secondary Outcome: Number of Participants Experiencing a Clinically Significant Episode of Urinary Retention
Description: as for outcome 18
Time Frame: up to 28 days or until discharge from the ICU (whichever is first)
Population: Participants with data collected. No participants were enrolled in the Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr) group.
Measure: Count of Participants; unit: Participants
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
Number analyzed (Participants) | 5 | 11 | 11 | 0
Participants | 1 | 2 | 1 |

23. Other Pre Specified Outcome: Average Daily Cornell Assessment of Pediatrics in Delirium (CAPD) Scores
Description: Estimate the incidence of intensive care unit delirium in children exposed to fentanyl and dexmedetomidine alone or in combination when receiving mechanical ventilation. (Measures of delirium). The CAPD scale goes from 0-4 and has 8 questions. All items scored as occurring never, rarely, sometimes, often, or always. Individual item scores are added for a sum total score.
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Maximum Daily CAPD Scores
Description: as for outcome 23
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Minimum Daily CAPD Scores
Description: as for outcome 23
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Average Daily Withdrawal Assessment Tool (WAT-1) Score
Description: Estimate the incidence of opioid withdrawal syndrome in children exposed to fentanyl and dexmedetomidine when administered alone or in combination when receiving mechanical ventilation. (Measures of withdrawal). WAT-1 scale is 0=no/none and 1=yes/moderate/severe. Total score is on a 0-12 scale where lower is better.
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Minimum Daily WAT-1 Score
Description: as for outcome 26
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Maximum Daily WAT-1 Score
Description: as for outcome 26
Time Frame: through day 7 of mechanical ventilation or initial extubation (whichever is first)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 28 days or until discharge from the ICU (whichever is first)
Description: No participants were enrolled in the Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr) group.
Arm/Group | Fen. SOC+Saline Placebo (Bolus+Infusion) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/12 | 0/12 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/12 | 1/12 | 0/0
Other Adverse Events (participants affected / at risk) | 4/6 | 9/12 | 8/12 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fen. SOC+Saline Placebo (Bolus+Infusion) (N=6) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) (N=12) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) (N=12) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr) (N=0)
General signs and symptoms NEC (General disorders) | 0 | 1 (1) | 0 | NA
Colitis (excl infective) (Gastrointestinal disorders) | 0 | 1 (1) | 0 | NA
Seizures and seizure disorder NEC (Nervous system disorders) | 0 | 0 | 1 (1) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fen. SOC+Saline Placebo (Bolus+Infusion) (N=6) | Fen. SOC+Dex.(.5mcg/kg + .25mcg/kg/hr) (N=12) | Fen. SOC+Dex.(.5mcg/kg + .5mcg/kg/hr) (N=12) | Fen. SOC+Dex.(.5mcg/kg + .75mcg/kg/hr) (N=0)
Anaesthetic and allied procedural complications (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA
Anxiety symptoms (Psychiatric disorders) | 0 | 1 | 0 | NA
Bladder and urethral symptoms (Renal and urinary disorders) | 1 | 2 | 1 | NA
Colitis (excl infective) (Gastrointestinal disorders) | 0 | 1 | 0 | NA
Conditions associated with abnormal gas exchange (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA
Encephalopathies NEC (Nervous system disorders) | 0 | 1 | 0 | NA
Febrile disorders (General disorders) | 2 | 0 | 1 | NA
General signs and symptoms NEC (General disorders) | 0 | 1 | 0 | NA
Heart rate and pulse investigations (Investigations) | 1 | 0 | 0 | NA
Hepatic failure and associated disorders (Hepatobiliary disorders) | 0 | 1 | 0 | NA
Laryngeal spasm, oedema and obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA
Magnesium metabolism disorders (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA
Nausea and vomiting symptoms (Gastrointestinal disorders) | 0 | 0 | 1 | NA
Parainfluenzae viral infections (Infections and infestations) | 1 | 0 | 0 | NA
Pneumothorax and pleural effusions NEC (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | NA
Protein metabolism disorders NEC (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA
Rate and rhythm disorders NEC (Cardiac disorders) | 2 | 5 | 5 | NA
Renal failure and impairment (Renal and urinary disorders) | 0 | 2 | 0 | NA
Respiratory tract and thoracic cavity procedural complications (Injury, poisoning and procedural complications) | 0 | 2 | 0 | NA
Seizures and seizure disorders NEC (Nervous system disorders) | 0 | 0 | 1 | NA
Stereotypies and automatisms (Psychiatric disorders) | 0 | 0 | 1 | NA
Tremor (excl congenital) (Nervous system disorders) | 0 | 0 | 1 | NA
Vascular hypotensive disorders (Vascular disorders) | 3 | 6 | 5 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT03938857/Prot_SAP_001.pdf
  • Informed Consent Form (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT03938857/ICF_000.pdf